CLINICAL TRIAL: NCT04039425
Title: Effects of Chemotherapy on the Concentration of Minerals in Hair
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Edward Bitok, Assistant Professor, Department of Nutrition and Dietitics, Loma Linda University
Other Study IDs: 5190216
Record Dates: First submitted 2019-07-25; First posted 2019-07-31 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cancer patient: * Recently diagnosed cancer stage 1, 2, or 3
  * Assigned to receive immunosuppressive chemotherapy treatment
  * Natural hair that has not been dyed or permed in the past 3 months
  Interventions: Procedure: Hair cut

INTERVENTIONS:
Procedure: Hair cut — Use only head hair. Cut samples of hair from back of head (see illustration). Cut hair as close to the scalp as possible. As each piece of hair is cut from the head, save only 3.7 square inches of hair closest to the scalp. According to the Doctors Data Lab, this amount is about enough hair to fill a tablespoon. Cut off and discard the rest. Place the saved hair on the scale. Keep cutting and adding hair to the scale until it tips. Hair collection will be about the weight of one to two paper clips (about 3800 strands). Remove the hair on the scale and put it in the plastic bag. Label the plastic bag with the patient's unique random identification and the date collected. Put the hair into the plastic bag, seal, and send to The Doctor's Data Lab.

SUMMARY:
The purpose of the investigator's graduate student research study is to investigate if there are significant changes in hair mineral levels in cancer patients undergoing chemotherapy.

DETAILED DESCRIPTION:
Visit 1 - Before the start of chemotherapy

* Complete a questionnaire about demographics, health, and diet.
* Weight and height will be measured.
* A small sample of the participant's hair will be collected from the back side of the head near the base of the neck. Only the hair in the first inch closest to the scalp will be included in the sample. This hair sample will weigh 0.25g to 1g, which is about the same weight as one to two regular paper clips.
* The participant will be given a food frequency questionnaire

Visit 2- Approximately 2 months after start of chemotherapy

* The participant will complete a questionnaire about their health and diet.
* weight and height will be measured
* A small sample of the participant's hair will be collected from the back side of the head near the base of the neck. Only the hair in the first inch closest to the scalp will be included in the sample. This hair sample will weigh 0.25g to 1g, which is about the same weight as one to two regular paper clips.
* The participant will be given a food frequency questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years and older
* Recently diagnosed cancer stage 1, 2, or 3
* Assigned to receive immunosuppressive chemotherapy treatment
* Natural hair that has not been dyed or permed in the past 3 months

Exclusion Criteria:

• Prior chemotherapy treatment for cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with any type of cancer, Stages 1, 2 or 3, assigned to receive immunosupressive chemotherapy treatment.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
hair mineral levels(ug/g) | change between visit 1(baseline/start of chemotherapy) and visit 2 (about 2 months after visit 1)
  Mineral levels such as calcium, magnesium, manganese, lead, iron, copper, cobalt, and chromium will be tested. All mineral levels are in ug/g.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Bitok, DrPH, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States